CLINICAL TRIAL: NCT03128333
Title: Effectiveness of Self-monitoring Physical Activity With a Smartphone Application and Physiotherapy Coaching in Cancer Patients: a Randomized Controlled Trial (SMART-COACH Trial)
Brief Title: Self-Monitoring Physical Activity With a Smartphone Application and Physiotherapy Coaching in Cancer Patients.
Acronym: SMART-COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201600902
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RunKeeper app + physiotherapy coaching (Experimental): Group A will use the RunKeeper app for half a year to self-monitor leisure-time PA. Besides, patients are requested to activate the 'training reminder' option in the RunKeeper app, which is all explained in a brief user's manual. In addition, patients will be educated about the health risks of a sedentary lifestyle, inactivity and (when applicable) other unhealthy lifestyle behaviors (e.g. unhealthy diet, overweight or obesity, sun exposure, alcohol intake). Benefits of a behavior change, becoming physically active and pursuing a healthy lifestyle will be explained by a trained physiotherapist who will also coach the patient during the PA program.
  Interventions: Other: RunKeeper app + physiotherapy coaching
- usual care (Other): In the UMCG, patients who receive cancer treatment or in surveillance after treatment are normally advised to live healthy, stay active, and to maintain their weight.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: RunKeeper app + physiotherapy coaching — RunKeeper app for half a year to self-monitor leisure-time PA.
  Arms: RunKeeper app + physiotherapy coaching
Other: Usual care — In the UMCG, patients who receive cancer treatment or in surveillance after treatment are normally advised to live healthy, stay active, and to maintain their weight.
  Arms: usual care

SUMMARY:
The aim of this study is to examine whether self-monitoring PA with the RunKeeper app with additional physiotherapy coaching is superior in improving patients' self-reported leisure-time PA compared with usual care in cancer patients after 12 weeks.

This is a single-center, prospective, two-armed, randomized controlled trial. Adult cancer patients and cancer survivors are randomized in one of the two study arms, (Group A) RunKeeper app + physiotherapy coaching or (Group B) usual care.

Patients assigned to the intervention group will be instructed to use the RunKeeper app for 12 weeks to self-monitor leisure-time PA. In addition, patients will be educated about the health risks of a sedentary lifestyle, inactivity and (when applicable) other unhealthy lifestyle behaviors (e.g. unhealthy diet, overweight or obesity, sun exposure, alcohol intake). Benefits of a behavior change, becoming physically active and pursuing a healthy lifestyle will be explained by a trained physiotherapist who will also coach the patient during the PA program. The biweekly physiotherapy coaching starts at baseline and will follow a structured sequence of strategies to change patients PA behavior which will contribute to the adoption of leisure-time PA in patients daily living, so the program will be optimally tailored to the patients capabilities and preferences.

The primary endpoint is to examine the effectiveness of the RunKeeper use with additional physiotherapy coaching in improving patients' leisure-time PA compared with usual care in cancer patients as measured by the PASE subscale leisure-time Sum Score at baseline, 6, 12 and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age diagnosed with cancer (regardless of type/taxonomy) at the medical oncology department, UMCG
* Patients undergoing cancer treatment or surveillance
* WHO-performance score ≤1
* Signed informed consent

Exclusion Criteria:

* Inability to read or understand the Dutch language
* Inability to handle or not in possession of a smartphone (iPhone ≥4 or Android phones)
* Active user of the RunKeeper app
* Severe cardiac (recent cardiovascular event) or psychiatric disease
* Patients following supervised oncologic rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
examine the effectiveness of the RunKeeper use with additional physiotherapy coaching | 6 months
  To examine the effectiveness of the RunKeeper use with additional physiotherapy coaching in improving patients' leisure-time PA compared with usual care in cancer patients as measured by the PASE subscale leisure-time Sum Score at baseline, 6, 12 and 26 weeks.

SECONDARY OUTCOMES:
investigate the improvement in the percentage of patients meeting the prescribed total weekly minutes of leisure-time PA | 6 months
  To investigate the improvement in the percentage of patients meeting the prescribed total weekly minutes of leisure-time PA with moderate to vigorous intensity corresponding to the NNGB as measured by accelerometry (ActiGraph GT3X-BT) at baseline, 12 and 26 weeks.
investigate the improvement in patients' weekly total minutes of leisure-time PA and sedentary time | 6 months
  To investigate the improvement in patients' weekly total minutes of leisure-time PA and sedentary time as measured by the PASE subscales leisure-time Total Minutes of PA and Sedentary Time at baseline, 6, 12 and 26 weeks.
examine the improvement in patients' health-related quality of life (HR-QoL) | 6 months
  To examine the improvement in patients' health-related quality of life (HR-QoL) as measured by the European Organization for Treatment of Cancer QoL (EORTC QLQ-C30) questionnaire at baseline, 12 and 26 weeks.
examine the improvement in patients' self-efficacy | 6 months
  To examine the improvement in patients' self-efficacy as measured by the Algemene Competentie Schaal (ALCOS) questionnaire at baseline, 12 and 26 weeks.
explore patients' PA Stage of Change | 6 months
  To explore patients' PA Stage of Change as measured by the Physician-based Assessment and Counseling for Exercise (PACE) questionnaire at baseline, 12 and 26 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: A. M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ormel HL, van Zutphen EH, van der Schoot GGF, Gietema JA, Walenkamp AME. Effects of self-monitoring physical activity with a smartphone application combined with physiotherapy coaching in patients with cancer: a randomised controlled trial (SMART-COACH trial). J Cancer Surviv. 2025 Jul 15. doi: 10.1007/s11764-025-01862-w. Online ahead of print. PMID 40665202